CLINICAL TRIAL: NCT06412978
Title: Post-Operative Cosmesis and Skin Closure Methods After Cesarean Section
Brief Title: Post-Operative Cesarean Section Cosmesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00109639
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cesarean Delivery
Keywords: cosmetic improvement; surgical correction; Cosmesis
MeSH Terms: interventions — glycolide E-caprolactone copolymer

STUDY DESIGN:
Intervention Model Description: trial comparing skin closure with absorbable subcuticular staples with subcuticular suture
Who Masked: Outcomes Assessor
Masking Description: Scars will be digitally photographed by study staff and scored by 2 independent judges. The judges will be blinded to the closure method at time of scar evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subcuticular absorbable polyglycolic acid (INSORB) staples (Active Comparator): Insorb absorbable staples are used for skin closure
  Interventions: Procedure: absorbable subcuticular polyglycolic acid staples (INSORB)
- subcuticular absorbable polyglecaprone suture (Monocryl) (Active Comparator): Monocryl absorbable staples are used for skin closure
  Interventions: Procedure: subcuticular, polyglecaprone suture (Monocryl)

INTERVENTIONS:
Procedure: absorbable subcuticular polyglycolic acid staples (INSORB) — Insorb absorbable staples are used for skin closure
  Other Names: INSORB
  Arms: subcuticular absorbable polyglycolic acid (INSORB) staples
Procedure: subcuticular, polyglecaprone suture (Monocryl) — Monocryl absorbable staples are used for skin closure
  Other Names: Monocryl
  Arms: subcuticular absorbable polyglecaprone suture (Monocryl)

SUMMARY:
Given the high numbers of cesarean deliveries being performed today, there has been interest in optimizing surgical techniques. Several recent reviews have summarized the evidence for various steps of cesarean delivery, but surprisingly in many cases there is little scientific evidence on which to base the choice of surgical technique.

DETAILED DESCRIPTION:
Cesarean delivery is the most common surgical procedure performed in the United States, with over 1 million procedures performed per year. Based on recent Center for Disease Control (CDC) National Vital Statistics Report (2021) 32.1% of all births in the United States were via cesarean delivery. Given the high numbers of cesarean deliveries being performed today, there has been interest in optimizing surgical techniques. Absorbable staples, made from a combination of polylactic and polyglycolic acid, are a relatively new option for skin closure at the time of surgery. This study is a randomized trial that will investigates two cesarean skin closure techniques-subcuticular, polyglecaprone suture (Monocryl), and absorbable subcuticular polyglycolic acid staples (INSORB)-to determine if one is associated with better scar cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44
* Any race
* Any parity
* Scheduled cesarean section
* Neuraxial analgesia

Exclusion Criteria:

* Non-English Speaking
* Incarcerated
* Maternal Connective Tissue Disorder
* Systemic maternal steroid use
* Three prior cesarean deliveries
* Body Mass Index (BMI) >40

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females requiring Cesarean Section
Enrollment: 52 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
scar cosmetic score | Week 6
  Scars will be digitally photographed by study staff and scored by 2 independent judges (attending Obstetricians) according to the SCAR scale validated by Kantor with scores ranging from 0 (best) to 15 (worst).

SECONDARY OUTCOMES:
Number of Wound complications | Week 6
  wound complications (infection, dehiscence, seroma, hematoma, skin and fat necrosis, skin and fascial dehiscence)
length of hospital stay | Week 6
  days spent in hospital
amount of in-hospital intravenous opiate analgesic use | Week 6
  amount of in-hospital intravenous opiate analgesic use
amount of in-hospital oral NSAID analgesic use | Week 6
  amount of in-hospital oral NSAID analgesic use
amount of in-hospital oral opiate analgesic use | Week 6
  amount of in-hospital oral opiate analgesic use
patient rated subjective pain score | Week 6
  patient rated subjective pain score (0-10 based on visual analog scale) - 100-mm visual analog scale (VAS) ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
patient's overall satisfaction with cosmesis scores | Week 6
  The Patient and Observer Scar Assessment Scale (POSASA) All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). Higher scores meaning more scarring

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Nitsche, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the participant data collected during the trial and after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose propose use of the data that has been approved by an Institutional Review Board
URL: https://ctulbert@wakehealth.edu